CLINICAL TRIAL: NCT06949371
Title: Investigation of the Effects of Chronotype Differences on Balance and Muscle Strength in Young Adults
Acronym: Chronotype
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7691; Istanbul Medipol University (Registry Identifier: Istanbul Medipol University Ethics Committee)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Chronotype
Keywords: Chronotype; muscle strength; balance; functionality

STUDY DESIGN:
Who Masked: Participant
Masking Description: participant are blind in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning chronotype group (Experimental): All assessment measurements determined for individuals with morning chronotype will be performed first at 09:00 in the morning and then again at 19:00 in the evening.
  Interventions: Other: Morning chronotype
- Evening chronotype group (Experimental): All assessment measurements determined for individuals with evening chronotype will be performed first at 09:00 in the morning and then again at 19:00 in the evening.
  Interventions: Other: Evening chronotype

INTERVENTIONS:
Other: Morning chronotype — All assessment measurements determined for individuals with morning chronotype will be performed first at 09:00 in the morning and then again at 19:00 in the evening. Muscle strength balance assessments performed in the morning and evening will be compared.
  Arms: Morning chronotype group
Other: Evening chronotype — All assessment measurements determined for individuals with evening chronotype will be performed first at 09:00 in the morning and then again at 19:00 in the evening. Muscle strength balance assessments performed in the morning and evening will be compared.
  Arms: Evening chronotype group

SUMMARY:
The aim of this study is to investigate the effects of chronotype differences on balance and muscle strength in young adults. Chronotypes of all participants will be determined using the Morningness-Eveningness Questionnaire. All assessment measurements determined for young adult individuals will be performed first at 09:00 in the morning and then again at 19:00 in the evening.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of chronotype differences on balance and muscle strength in young adults. Inclusion criteria are being between 45-65 years old, not having any neurological or orthopedic disorders, not having a vestibular disease that causes balance problems. Exclusion criteria are trauma history, anatomical deformities and skeletal system fractures, having a previous injury, and the presence of pain that will prevent participation in the tests. Chronotypes of all participants will be determined using the Morningness-Eveningness Questionnaire. All assessment measurements determined for young adult individuals will be performed first at 09:00 in the morning and then again at 19:00 in the evening. Muscle strength and balance assessments made in the morning and evening will be compared. Chronotypes of the participants will be evaluated with the Morningness-Eveningness Questionnaire, their balance will be evaluated with the One-Legged Standing Test, lower extremity muscle strength with a myometer, and their functionality will be evaluated with the Timed Stand-Up-Sit Test and the 30-Second Sit-Up Test.

ELIGIBILITY:
Inclusion Criteria:

* being between 45-65,
* not having any neurological or orthopedic disorder,
* not having a vestibular disease that causes balance problems.

Exclusion Criteria:

* trauma history,
* anatomical deformities and skeletal system fractures,
* having a previous injury and the presence of pain that would prevent participation in the tests.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Morningness-Eveningness Questionnaire | 20 minutes
  A questionnaire form that determines morningness and eveningness types will be used to subjectively evaluate circadian rhythm. defi - nitely morning type (70-86), moderately morning type (59-69), neither type (42-58), moderately evening type (31-41), and defi nitely evening type (16-30).
Single-leg standing test | 20 minutes
  This test measures a person's standing ability and balance.
Muscle strength test | 20 minutes
  Myometry will be used to objectively measure the strength of the quadriceps and hamstring muscles. Myometry is an evaluation method that objectively evaluates muscle strength and provides more sensitive results than manual muscle testing.
Timed up and go testTest: | 20 minutes
  A simple screening test that provides a sensitive and specific measure of fall risk and balance in older adults.
30 Second Sit-to-Stand Test | 20 minutes
  A test that evaluates the participant's sit-to-stand activity, lower extremity muscle strength and balance status.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Assoc. Prof., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We can share IPD when it isi necessary.

REFERENCES:
- [Result] Facer-Childs ER, Boiling S, Balanos GM. The effects of time of day and chronotype on cognitive and physical performance in healthy volunteers. Sports Med Open. 2018 Oct 24;4(1):47. doi: 10.1186/s40798-018-0162-z. PMID 30357501
- See also: The effects of time of day and chronotype on cognitive and physical performance in healthy volunteers — https://pmc.ncbi.nlm.nih.gov/articles/PMC6200828/